CLINICAL TRIAL: NCT02563028
Title: A Novel Method for Capturing the Visual Evoked Potential (VEP) During Single-Level Lumbar Spine Decompression/Fusion Under Total Intravenous Anesthesia (TIVA)
Brief Title: A Novel Method for Capturing the Visual Evoked Potential During Spine Surgery Under Total Intravenous Anesthesia
Acronym: VEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-272
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Evoked Potentials, Visual
Keywords: Visual Evoked Potentials; Microdiscectomy; SightSaver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SightSaver Visual Stimulator (Experimental): A SightSaver Visual Stimulator mask will be applied during surgery. Baseline VEPs will be recorded prior to prone positioning. At the end of surgery, after supine positioning, the SightSaver Visual Stimulator mask will be removed and discarded.
  Interventions: Device: SightSaver Visual Stimulator

INTERVENTIONS:
Device: SightSaver Visual Stimulator — Evoked response photic stimulator

SUMMARY:
Spine surgery in the prone position (which involves lying face down) is associated with various visual changes, ranging from temporary changes in acuity (or sharpness) to permanent blindness. Known risk factors include low blood count (anemia) and long surgical times in the prone position under general anesthesia. While blindness is a rare outcome of this surgery, it is devastating and incompletely prevented by controlling known risk factors. Thus, improved monitoring and detection of visual injury during surgery is necessary. The purpose of this study is to determine whether a novel, non-invasive monitoring device can reliably record visual responses during spine surgery. The first phase of this study is completed and involved patients undergoing microdiscectomy surgery. The second phase of this study involves patients undergoing single-level lumbar spine decompression/fusion surgery.

DETAILED DESCRIPTION:
Spine surgery is associated with a variety of post-operative visual complications, ranging from mild, transient deficits in acuity to full visual loss. Known risk factors for visual loss include anemia, hypotension, and long surgical times in the prone position under general anesthesia. Despite recognition and control of risk factors, the prevalence of visual loss after prone spine surgery is estimated at approximately 0.1-1% . The pathophysiology of visual loss most often reflects posterior ischemic optic neuropathy, but anterior ischemic optic neuropathy and posterior reversible encephalopathy syndrome have also been described.

These reports suggest that the entire pathway from retina to visual cortex is vulnerable to injuries causing post-operative visual deficits. The potential for severe injury during spine surgery mandates improved detection of evolving optic tract injury during prone spine surgery.

Theoretically, the flash visual evoked potential (VEP) represents a useful intraoperative tool to monitor global visual system function. However, its application to spine surgery has been limited due to challenges in acquiring and interpreting signals intraoperatively. Several devices for intraoperative VEP-recording have been described . However, most of these have been trialed with patients in the supine or beach chair position, undergoing neurosurgical procedures. Goggle or eyepatch-designed devices have the potential to move during surgery, changing the relationship between the goggle and globe. The goggle itself may potentially compress the globe, producing inconsistent illumination to the retina or causing mechanical injury. These are particular liabilities during changes in position from supine to prone, as is required for many spine surgeries. Additionally, VEPs are extremely variable and exquisitely sensitive to anesthetics- particularly inhaled agents. Consistent with this, intravenous (rather than inhaled) agents have been associated with successful intraoperative VEP monitoring patients, particularly in patients without baseline visual impairment. Nonetheless, there are multiple reports in the literature showing poor correlation/prediction of postoperative visual status by intraoperative VEP measurements. A novel technology for capturing VEPs has recently been developed and may address several of the liabilities described above. The device is constructed from soft foam padding in a "ski mask" design, which we hypothesize may add a measure of protection to the eyes compared to traditional VEP goggles or patches. This design may also provide stability during changes in patient positioning from supine to prone. The front of the mask consists of an opaque circuit board with six bright light emitting diodes positioned in front of each eye, allowing illumination of the retina through closed, protected eyes. Opaque foam separates right and left sides of the mask, allowing each eye to be stimulated individually. To date, the mask has not been tested for sensitivity to elicit and record VEPs in patients under anesthesia. In this pilot study, we tested the feasibility of using the mask during prone spine surgery. Specifically, we asked if VEPs can be detected throughout spine surgeries of varying complexity and duration, whether the signals change with changes in patient positioning and anesthetic conditions, and whether the mask was associated with any adverse effects. Here we show that intraoperative VEPs can be recorded throughout spine surgery using this device. We also describe effects of several anesthetic agents on VEP stability, and ask if there is any qualitative relationship between changes in VEPs and SSEPs recorded simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting for single-level microdiscectomy (first phase only)
* Any patient presenting for single-level lumbar spine decompression/fusion (second phase only)
* Any patient suitable for total intravenous anesthesia (TIVA)
* Age >18

Exclusion Criteria:

* Neurologic or demyelinating disease expected to be associated with impaired VEPs
* Eye disease, including blindness, glaucoma, macular degeneration, diabetic retinopathy, or conditions expected to be associated with impaired VEPs
* Patients with a known history of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Beckman, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Result] Soffin EM, Emerson RG, Cheng J, Mercado K, Smith K, Beckman JD. A pilot study to record visual evoked potentials during prone spine surgery using the SightSaver photic visual stimulator. J Clin Monit Comput. 2018 Oct;32(5):889-895. doi: 10.1007/s10877-017-0092-1. Epub 2017 Dec 20. PMID 29264762

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraoperative Monitoring Device: In this study, the FDA-cleared, non-invasive mask called SightSaverTM Visual Stimulator is used as an additional monitor to identify potential changes in the visual system during surgery
Period: Overall Study
Arm/Group | Intraoperative Monitoring Device
Started | 20
Completed | 18
Not Completed | 2
Not completed — Lack of equipment | 1
Not completed — Unable to elicit VEP post induction | 1

BASELINE CHARACTERISTICS:
Population: Any patient presenting for microdiscectomy, single level lumbar spine decompression/fusion, or multilevel posterior spine fusion
Groups:
- Evoked Response Photic Stimulator: Arms
  Assigned Interventions
  Experimental: SightSaver Visual Stimulator
  A SightSaver Visual Stimulator mask will be applied during surgery. Baseline VEPs will be recorded prior to prone positioning. At the end of surgery, after supine positioning, the SightSaver Visual Stimulator mask will be removed and discarded.
  Device: SightSaver Visual Stimulator
  Evoked response photic stimulator
Arm/Group | Evoked Response Photic Stimulator
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of VEPs
Description: The primary outcome will be the presence of VEPs during spine surgery. This outcome will be measured in realtime, intraoperatively. Outcome measure: Visual evoked potential morphology, varying in amplitude (µV) and latency.
Time Frame: Duration of surgery (approximately 3 hours)
Population: Patients >18 years old who underwent posterior spine surgery with general anesthesia were enrolled. Surgeries were microdiscectomy or instrumented fusion, irrespective of surgical type or patient position (supine or prone).
Measure: Count of Participants; unit: Participants
Arm/Group | SightSaver Visual Stimulator
Number analyzed (Participants) | 18
Participants | 18

2. Secondary Outcome: Number of Participants With Change in VEP Signal Strength
Description: Number of participants with change in VEP signal strength. This outcome will be measured in realtime, intraoperatively.
Time Frame: Duration of surgery (approximately 3 hours)
Population: Patients who were >18 years old and were undergoing posterior spine surgery with general anesthesia were approached for the study. Eligible surgeries were microdiscectomy or instrumented fusion (lumbar, thoracic, or thoraco-lumbar). There were no restrictions on the number of surgical levels for inclusion in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SightSaver Visual Stimulator
Number analyzed (Participants) | 18
Participants | 18

3. Secondary Outcome: Correlation of Change in VEPs With Identifiable Intraoperative Event
Description: Whether changes in VEPs vary with any identifiable intraoperative change in patient condition (including hypotension, hypertension, tachycardia, bradycardia, arrhythmias, oxygen saturation, CO2 level, hypothermia and hyperthermia), surgical event (including sudden or ongoing hemorrhage, neurological injury), or anesthetic change (including increasing/decreasing doses of anesthetics, depth of anesthesia and use of vasoactive drugs). This outcome will be measured in realtime, intraoperatively. Number of participants with change in VEPs associated with increases or decreases of isoflurane and nitrous oxide are reported.
Time Frame: Duration of surgery (approximately 3 hours)
Population: Correlation of change in VEPs was qualitatively examined in 18 patients, but not systematically quantified.
Measure: Number; unit: participants
Arm/Group | SightSaver Visual Stimulator
Number analyzed (Participants) | 18
participants | 18

4. Secondary Outcome: Number of Participants With Intolerance to the SightSaver Visual Stimulator
Description: Whether the SightSaverTM Visual Stimulator is well tolerated by patients. This outcome will be assessed in the PACU will comprise a clinical exam of the periorbital structures and a patient questionnaire
Time Frame: Postoperatively, after recovery from anesthesia (approximately 3 hours after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | SightSaver Visual Stimulator
Number analyzed (Participants) | 18
Participants | 1

ADVERSE EVENTS:
Time Frame: Patients were followed up until Post Anesthesia Care Unit (PACU) by the anesthesiologists. A survey was filled out by the anesthesiologists to assure the wellness of the patient. Up to 24 hours after surgery.
Description: This is a pilot study (non-invasive) where there was no treatment involved thus there were no interventions.
  There was a 5% incidence of Adverse Event.
Groups:
- SightSaver Visual Stimulator: A SightSaver Visual Stimulator mask will be applied during surgery. Baseline VEPs will be recorded prior to prone positioning. At the end of surgery, after supine positioning, the SightSaver Visual Stimulator mask will be removed and discarded.
  SightSaver Visual Stimulator: Evoked response photic stimulator
  Adverse event total: 0/20 0%
Arm/Group | SightSaver Visual Stimulator
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SightSaver Visual Stimulator (N=20)
Minor periorbital skin irritation. (Skin and subcutaneous tissue disorders) | 1 (1) — One patient reported minor periorbital skin irritation, which was unaccompanied by physical findings, and resolved fully prior to discharge from the PACU.

LIMITATIONS AND CAVEATS:
Twenty patients were enrolled but only 18 were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No